CLINICAL TRIAL: NCT04645108
Title: Randomized, Parallel Trial of Overweight Men and Women Using a Coached or Non-Coached Weight Loss Intervention
Brief Title: Coached or Non-Coached Weight Loss Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Noom Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00046922
Record Dates: First submitted 2020-10-28; First posted 2020-11-27 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Obesity; Behavior, Health; Behavior, Eating; Weight Loss; Overweight and Obesity; Self Efficacy
MeSH Terms: conditions — Obesity; Health Behavior; Feeding Behavior; Weight Loss; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coached (Experimental)
  Interventions: Behavioral: Noom Healthy Weight; mobile behavior change program for weight loss with 1:1 coaching
- No Coach (Active Comparator)
  Interventions: Behavioral: Noom Healthy Weight; mobile behavior change program for weight loss

INTERVENTIONS:
Behavioral: Noom Healthy Weight; mobile behavior change program for weight loss with 1:1 coaching — The intervention consists of a curriculum, provided through daily articles that users are encouraged to read; logging features for weight, meals, and physical activity; in-app groups; and a virtual coach, who will communicate with participants via in-app messaging. During the first week of the study, participants will be introduced to the program, the Noom app, and their coach.
  Coaches will use a secure dashboard to monitor patient progress, which is used to increase engagement and motivation. Participants are encouraged to log their weight and physical activity on a weekly basis, and meals daily.
  Arms: Coached
Behavioral: Noom Healthy Weight; mobile behavior change program for weight loss — The intervention consists of a curriculum, provided through daily articles that users are encouraged to read; logging features for weight, meals, and physical activity. During the first week of the study, participants will be introduced to the program, and the Noom app.
  Arms: No Coach

SUMMARY:
To evaluate the effect of one-on-one coaching in the Noom Healthy Weight Program, a digital behavior change, weight loss intervention, compared to the same program with no coaching, as well as influential factors.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and provide informed consent
* 18-65 years old
* Self-report of good health (physical and mental)
* Not diagnosed with diabetes
* Overweight or obesity (BMI ≥ 27)
* Able to meet our criteria of adherence to the program (at least 1 engagement per week on one of the following: logged exercise, logged meals, steps, weigh-ins, coach messages, read articles, and days with at least one weigh-in.) For females
* Not 6 months postpartum
* Not planning to become pregnant in the next 5 months.

Exclusion Criteria:

* Inability or unwillingness of a participant to give written informed consent
* Currently pregnant or ≤ 6 months postpartum
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the quality of the data E.g., evidence of an eating disorder, major chronic condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Weight | 4 months
  Self reported
Self reported in app engagement measures | 4 months
  self reported and automatically logged

SECONDARY OUTCOMES:
Quality of Life Via SF-12 | 4 months
  Self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure
Eating Behavior via the Dutch Eating Behavior Questionnaire | 4 months
  The Dutch Eating Behavior Questionnaire (DEBQ) assesses the structure of an individual's eating behavior. the DEBQ contains separate scales for emotional, external, and restrained eating behavior.
Resilience via Devereux Adult Resilience Survey | 4 months
  Provides insights into personal strengths
Self Efficacy via General Self-Efficacy Scale | 4 months
  The scale was created to assess a general sense of perceived self-efficacy with the aim in mind to predict coping with daily hassles as well as adaptation after experiencing all kinds of stressful life events.
Linguistic Features via Linguistic Inquiry Word Count (LIWC) | 16 weeks
  LIWC-derived linguistic analysis of emotional tone taken from from expressively written text following a writing task prompt

CONTACTS AND LOCATIONS:
Locations (1):
- Noom, Inc, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No